CLINICAL TRIAL: NCT01199822
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetic Profiles of IMC-3G3 Administered in a 2-week, or 3-week Schedule to Japanese Patients With Advanced Solid Tumors
Brief Title: Study of the Safety and Pharmacokinetics of Olaratumab (IMC-3G3) in Japanese Participants With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13940; CP15-0907 (Other: ImClone, LLC); I5B-IE-JGDF (Other: Eli Lilly and Company); 21-3720 (Other: PMDA (MoH) in Japan)
Record Dates: First submitted 2010-09-08; First posted 2010-09-13 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Malignancy; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — olaratumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Olaratumab (Experimental)
  Interventions: Biological: Olaratumab

INTERVENTIONS:
Biological: Olaratumab — Cohort 1 10 milligrams/kilogram (mg/kg) intravenously (IV) administered on Days 1 and 8, every 3 weeks; Cohort 2 20 mg/kg IV administered every 2 weeks; Cohort 3 15 mg/kg IV administered on Days 1 and 8, every 3 weeks
  Other Names: IMC-3G3; LY3012207

SUMMARY:
Participants in this single-center, open-label, dose-escalation, Phase 1 study will initially receive intravenous (IV) olaratumab once every 2 weeks or on Days 1 and 8 every 3 weeks for 6 weeks (one cycle). After the first cycle, participants experiencing an overall response of complete response (CR), partial response (PR), or stable disease (SD) will continue to receive olaratumab at their cohort dose and schedule until there is evidence of progressive disease (PD), or until other withdrawal criteria are met.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor that has been histopathologically or cytologically documented
* Advanced primary or recurrent solid tumor participants who has not responded to standard therapy or for whom no standard therapy is available
* Measurable or nonmeasurable lesions
* An Eastern Cooperative Oncology Group Performance Status score of 0-1
* Able to provide informed consent
* Has a life expectancy of >3 months
* Adequate hematologic function
* Adequate hepatic function
* Has adequate renal function
* Agrees to use adequate contraception for the duration of study participation and for at least 12 weeks after the last dose of study therapy
* Adequate recovery from recent surgery, chemotherapy, and radiation therapy (including palliative radiation therapy). At least 28 days (6 weeks for nitrosoureas or mitomycin C) must have elapsed from major surgery, prior chemotherapy, prior treatment with an investigational agent or device, or prior radiation therapy. For treatment with non-approved monoclonal antibodies, a minimum of 8 weeks must have elapsed
* Is willing to comply with study procedures until the End-of-Therapy visit

Exclusion Criteria:

* Received chemotherapy or therapeutic radiotherapy within 28 days (6 weeks for nitrosoureas or mitomycin C) prior to entering the study, or has ongoing side effects ≥ Grade 2 due to agents administered more than 28 days earlier
* Has undergone major surgery [example (e.g.), laparotomy, thoracotomy, removal of organ(s)] within 28 days prior to study entry
* Elective or planned surgery to be conducted during the trial
* Documented and/or symptomatic brain or leptomeningeal metastases (participants who are clinically stable [no symptoms during the 4 weeks prior to study entry] with an assessment that no further treatment [radiation, surgical excision, or administration of steroids] is required are permitted to enter the study)
* Uncontrolled intercurrent illness including, but not limited to:

  * Active infection requiring systemic antibiotic treatment excluding oral administration [≥Grade 3 National Cancer Institute - Common Terminology Criteria for Adverse Events [NCI-CTCAE Version (v) 4.02)]
  * Congestive heart failure (Class III or IV per the New York Heart Association classification for heart disease)
  * Angina pectoris, angioplasty, stenting, or myocardial infarction within 6 months
  * Uncontrolled hypertension [systolic blood pressure >150 millimeters of mercury (mm Hg), diastolic blood pressure >95 mm Hg]
  * Cardiac arrhythmia requiring treatment (NCI-CTCAE v4.02, or asymptomatic sustained ventricular tachycardia
  * Peripheral neuropathy of any etiology ≥Grade 2 (NCI-CTCAE v4.02); or
  * Any other serious uncontrolled medical disorder(s) in the opinion of the investigator
* Participated in clinical studies of non-approved experimental agents or procedures within 4 weeks prior to study for small molecules, or 8 weeks prior to study entry for non-approved monoclonal antibodies
* Received any previous treatment with agents targeting the platelet-derived growth factor (PDGF) or platelet-derived growth factor receptor (PDGFR), approved or non-approved
* Known allergy to any of the treatment components (IMC-3G3, histidine, glycine, sodium chloride, mannitol, or polysorbate)
* If female, is pregnant (confirmed by urine or serum pregnancy test) or lactating
* Known alcohol or drug dependency
* Hepatitis B virus (HBV) antigen-, hepatitis C virus (HCV) antibody-, or human immunodeficiency (HIV) antibody-positive [asymptomatic healthy carriers with detectable HBV-Deoxyribonucleic acid (DNA), HCV-Ribonucleic acid (RNA) may be enrolled into the trial]
* Assessed as inadequate for the study by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- ImClone Investigational Site, Kashiwa, Chiba, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: There were 3 cohorts and enrollment into the next cohort did not occur until all participants in the previous cohort completed 1 cycle of treatment or discontinued due to dose-limiting toxicity (DLT). Participants who completed Cycle 1 or had DLT during Cycle 1 are considered having completed study.
Groups:
- 10 mg/kg Olaratumab (IMC-3G3): 10 milligrams/kilogram (mg/kg) olaratumab intravenously (IV) administered on Days 1 and 8, every 3 weeks (6-week cycle). Cycles repeated until there was evidence of progressive disease (PD), or until other withdrawal criteria were met.
- 20 mg/kg Olaratumab: 20 mg/kg olaratumab IV administered on Day 1 every 2 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met.
- 15 mg/kg Olaratumab: 15 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met.
Period: Overall Study
Arm/Group | 10 mg/kg Olaratumab (IMC-3G3) | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Started | 3 | 7 | 6
Received at Least 1 Dose of Study Drug | 3 | 7 | 6
Completed | 3 | 6 | 6
Not Completed | 0 | 1 | 0
Not completed — Investigator discontinued therapy | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 dose of study drug.
Groups:
- 10 mg/kg Olaratumab: 10 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met.
- Total: Total of all reporting groups
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab | Total
Number analyzed (Participants) | 3 | 7 | 6 | 16
Age, Customized [Number; unit: participants]
  20 - <65 Years | 1 | 6 | 4 | 11
  ≥65 Years | 2 | 1 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 4 | 6
  Male | 3 | 5 | 2 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 7 | 6 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Japan | 3 | 7 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: Data presented are the number of participants who experienced AEs of any grade and AEs of Grade ≥3 as determined by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 4.02. A summary of serious adverse events (SAEs) and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose to study completion up to 5.6 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 3 | 7 | 6
participants
  AE of Any Grade | 3 | 7 | 6
  AE of Grade ≥3 | 1 | 1 | 0

2. Primary Outcome: Number of Participants With SAEs
Description: A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: First dose to study completion up to 5.6 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 3 | 7 | 6
participants | 0 | 1 | 0

3. Primary Outcome: Number of Participants With a Dose- Limiting Toxicity (DLT) in Cycle 1
Description: A DLT is defined as 1 of the following events, if considered by the investigator to be definitely, probably, or possibly related to olaratumab: NCI-CTCAE v4.02 Grade 4 neutropenia lasting >7 days; NCI-CTCAE v4.02 Grade ≥3 thrombocytopenia with signs of bleeding or requiring platelet transfusions; NCI-CTCAE v4.02 Grade ≥3 neutropenia associated with fever; NCI-CTCAE v4.02 Grade 3 or 4 nonhematologic toxicity, excluding electrolyte abnormality; NCI-CTCAE v4.02 Grade ≥3 skin toxicity despite best preemptive and supportive care; and/or NCI-CTCAE v4.02 Grade ≥3 diarrhea, nausea, or vomiting despite best preemptive and supportive care.
Time Frame: First dose through Cycle 1 (6 weeks/cycle)
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Groups:
- 10 mg/kg Olaratumab: 10 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle) during Cycle 1.
- 20 mg/kg Olaratumab: 20 mg/kg olaratumab IV administered on Day 1 every 2 weeks (6-week cycle) during Cycle 1.
- 15 mg/kg Olaratumab: 15 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle) during Cycle 1.
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 3 | 7 | 6
participants | 0 | 0 | 0

4. Primary Outcome: Maximum Concentration (Cmax) of Olaratumab Following Multiple Doses
Time Frame: Cycle 2: Pre-dose and up to 336 hours post-dose
Population: All participants who received study drug and had pharmacokinetic (PK) data available to calculate Cmax. Due to the limited data, Cmax is not representative of the study population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/mL)
Groups:
- 10 mg/kg Olaratumab: 10 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle) during Cycles 1 and 2.
- 20 mg/kg Olaratumab: 20 mg/kg olaratumab IV administered on Day 1 every 2 weeks (6-week cycle) during Cycles 1 and 2.
- 15 mg/kg Olaratumab: 15 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle) during Cycles 1 and 2.
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 2 | 3 | 1
micrograms/milliliter (µg/mL) | 603 (NA) — 2 participants were analyzed; therefore arithmetic mean was calculated and geometric coefficient of variation was not calculated. | 1160 (91) | 921 (NA) — 1 participant was analyzed; therefore actual value was presented and geometric coefficient of variation was not calculated.

5. Secondary Outcome: Area Under the Concentration of Olaratumab Versus Time Curve During One Dosing Interval (AUCτ) Following Multiple Doses
Time Frame: Cycle 2: Pre-dose and up to 336 hours post-dose
Population: All participants who received study drug and had PK data available to calculate AUCτ. Zero participants were analyzed for groups of 10 mg/kg IMC-3G3 and 15 mg/kg IMC-3G3 because of insufficient amount of samples collected. Due to the limited data, AUCτ is not representative of the study population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms*hours/milliliter (µg*h/mL)
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 0 | 3 | 0
micrograms*hours/milliliter (µg*h/mL) |  | 123000 (29) |

6. Secondary Outcome: Terminal Elimination Half-Life (t1/2) of Olaratumab
Description: t1/2 is the time it takes for the drug concentration in serum to decrease to half the value observed at the beginning of the time period.
Time Frame: Cycle 2: Pre-dose and up to 336 hours post-dose
Population: All participants who received study drug and had PK data available to calculate t1/2. Due to limited data and the relatively short duration of sample collection, t1/2 is not representative of the study population.
Measure: Geometric Mean (Full Range); unit: days
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 2 | 3 | 1
days | NA [4.06 to 7.33] — 2 participants were analyzed; therefore geometric mean was not calculated. | 7.33 [5.42 to 8.83] | 8.25 [NA to NA] — 1 participant was analyzed; therefore actual value was presented and range was not provided.

7. Secondary Outcome: Clearance of Olaratumab at Steady State (CLss)
Description: CLss is the volume of plasma (or blood) from which the drug is completely removed, or cleared, in a given time at steady-state.
Time Frame: Cycle 2: Pre-dose and up to 336 hours post-dose
Population: All participants who received study drug and had PK data available to calculate CLss. Zero participants were analyzed for groups of 10 mg/kg IMC-3G3 and 15 mg/kg IMC-3G3 because of insufficient amount of samples collected. Due to limited data, CLss is not representative of the study population.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliters/hour/kilogram (mL/h/kg)
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 0 | 3 | 0
milliliters/hour/kilogram (mL/h/kg) |  | 0.163 (29) |

8. Secondary Outcome: Volume of Distribution at Steady State (Vss)
Time Frame: Cycle 2: Pre-dose and up to 336 hours post-dose
Population: Zero participants were analyzed because of insufficient amount of samples collected.
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Serum Anti-Olaratumab Antibody Assessment (Immunogenicity)
Description: Participants with Treatment Emergent (TE) anti-olaratumab antibodies were participants with a 4-fold increase (2 dilutions) increase over a positive baseline antibody titer or for a negative baseline titer, a participant with an increase from the baseline to a level of 1:20.
Time Frame: First dose to study completion up to 5.6 months
Population: All participants who received at least one dose of study drug and had evaluable baseline and evaluable post-baseline antibody data.
Measure: Number; unit: participants
Groups:
- Olaratumab: 10 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met. 20 mg/kg olaratumab IV administered on Day 1 every 2 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met. 15 mg/kg olaratumab IV administered on Days 1 and 8, every 3 weeks (6-week cycle). Cycles repeated until there was evidence of PD, or until other withdrawal criteria were met.
Arm/Group | Olaratumab
Number analyzed (Participants) | 15
participants | 0

10. Secondary Outcome: Number of Participants With Treatment Related AEs
Description: Data presented are the number of participants who experienced a treatment related AE of any grade.
Time Frame: First dose to study completion up to 5.6 months
Population: All enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Number analyzed (Participants) | 3 | 7 | 6
participants
  Any treatment related AE | 1 | 6 | 1
  Anaemia | 0 | 1 | 0
  Leukopenia | 0 | 1 | 0
  Diarrhoea | 0 | 1 | 0
  Fatigue | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 2 | 0
  Fibrin D dimer increased | 0 | 1 | 0
  Hyperglycaemia | 0 | 1 | 0
  Tumour haemorrhage | 0 | 1 | 0
  Proteinuria | 0 | 3 | 1
  Cough | 1 | 0 | 0
  Dermatitis | 0 | 0 | 1
  Rash | 0 | 1 | 0
  Hypertension | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | 10 mg/kg Olaratumab | 20 mg/kg Olaratumab | 15 mg/kg Olaratumab
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/7 | 0/6
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10 mg/kg Olaratumab (N=3) | 20 mg/kg Olaratumab (N=7) | 15 mg/kg Olaratumab (N=6)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10 mg/kg Olaratumab (N=3) | 20 mg/kg Olaratumab (N=7) | 15 mg/kg Olaratumab (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (2) | 1 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (5) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 0 (0)
Fibrin D dimer increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (4)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (4)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Proteinuria (Renal and urinary disorders) | 0 (0) | 3 (3) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0/0 (0) | 1/2 (1) | 0/4 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.